CLINICAL TRIAL: NCT06926829
Title: A Phase 3, Multicenter, Open-label, Uncontrolled, Long-term Trial to Evaluate the Safety and Efficacy of Long-term Administration of EB-1020 Once Daily QD XR Capsules in Adults With Attention-deficit/Hyperactivity Disorder
Brief Title: A Long-term Trial of EB-1020 in Adult Patients With ADHD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 405-102-00113
Record Dates: First submitted 2025-04-11; First posted 2025-04-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EB-1020 (QD XR Capsules) 164.4 mg (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) 164.4 mg
- EB-1020 (QD XR Capsules) 328.8 mg (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) 328.8 mg

INTERVENTIONS:
Drug: EB-1020 (Centanafadine) 164.4 mg — 164.4 mg, capsule, oral, once daily, for 52 weeks
  Arms: EB-1020 (QD XR Capsules) 164.4 mg
Drug: EB-1020 (Centanafadine) 328.8 mg — 328.8 mg, capsule, oral, once daily, for 52 weeks
  Arms: EB-1020 (QD XR Capsules) 328.8 mg

SUMMARY:
The purpose of this study is to evaluate the safety of long-term administration of mainly high doses of EB-1020 over 52 weeks in patients who have completed the double-blind trial (405-102-00112) conducted in Japan

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the treatment period andfollow-up period in the preceding double-blind parent Trial (Trial 405-102-00112) and did not meet the criteria for discontinuation of the investigational medicinal product (IMP).
* Participants who have not been found to have major problems with trial requirements, such as compliance with the IMP, in the preceding double-blind parent trial.

Exclusion Criteria:

* Participants who are pregnant or breastfeeding or test positive for pregnancy on baseline visit.
* Participants who started prohibited concomitant medications/therapies for ADHD or other comorbidities at the end of the follow-up period of the preceding trial, or participants for whom starting treatment is deemed beneficial.
* Participants who have a significant risk of committing suicide in the opinion of the investigator or subinvestigator, or based on the following evidence:

  * Active suicidal ideation as evidenced by an answer of "yes" on Questions 4 or 5 on the section of suicidal ideation on the since last visit version of the Columbia-Suicide Severity Rating Scale (C-SSRS) in the preceding double-blind parent trial or
  * Reported suicidal behavior
* Participants who were found to have serious or severe adverse events that were judged to be related to the IMP in the preceding double-blind parent trial.
* Participants who test positive for drugs or alcohol in a urine test on baseline visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Experiencing Treatment-Emergent Adverse Events (TEAEs) | Baseline, week52
  An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with an onset date on or after the first dose of IMP. They are all adverse events that started after the start of centanafadine; or if the event was continuous from baseline and was worsening, serious, study drug-related, or resulted in death, discontinuation, interruption or reduction of study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Maynds Tower Mental Clinic, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.